CLINICAL TRIAL: NCT00742612
Title: A Study of the Effect of ARC1779 Injection on Cerebral Microembolism in Patients Undergoing Carotid Endarterectomy
Brief Title: Effect of ARC1779 on Cerebral Microembolism in Patients Undergoing Carotid Endarterectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment slower than expected
Sponsor: Archemix Corp. (Industry)
Collaborators: St George's, University of London (Other)
Responsible Party: James Gilbert, MD./Chief Medical Officer, Archemix Corp.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARC1779-008
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2009-07

CONDITIONS: Intracranial Embolism; Cerebral Thromboembolism; Carotid Stenosis
Keywords: Carotid Endarterectomy; von Willebrand Factor; Microembolic Signal
MeSH Terms: conditions — Intracranial Embolism; Carotid Stenosis | interventions — ARC 1779; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): ARC1779 Injection
  Interventions: Drug: ARC1779 Injection
- 2 (Placebo Comparator): Placebo (normal saline)
  Interventions: Drug: Placebo (normal saline)

INTERVENTIONS:
Drug: ARC1779 Injection — Study drug treatment will be initiated 1 hour prior to the induction of anesthesia with a loading dose given over 1 hour in 3 successively increasing, 20-minute step infusions. The ARC1779 treatment group will be dosed to achieve a target ARC1779 steady-state plasma concentration of 3 Ug/mL, using a loading dose infusion sequence of 0.0015 mg/kg/min for 20 minutes, 0.003 mg/kg/min for the next 20 minutes, and then 0.006 mg/kg/min for the final 20 minutes; thereafter, their maintenance infusion rate is to be 0.0006 mg/kg/min.
  Arms: 1
Drug: Placebo (normal saline) — Study drug treatment will be initiated 1 hour prior to the induction of anesthesia with a loading dose given over 1 hour in 3 successively increasing, 20-minute step infusions. The placebo group will be dosed to a steady-state plasma concentration using a loading dose infusion sequence of 0.0015 mg/kg/min for 20 minutes, 0.003 mg/kg/min for the next 20 minutes, and then 0.006 mg/kg/min for the final 20 minutes; thereafter, their maintenance infusion rate is to be 0.0006 mg/kg/min.
  Arms: 2

SUMMARY:
The purpose of this study is to determine, in patients undergoing carotid endarterectomy, the effect of ARC1779 Injection on the number of microembolic signals detected by transcranial Doppler immediately after surgery. This study will also evaluate the safety of ARC1779 Injection with respect to bleeding risk in patients in the peri-operative (during surgery) period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients;
* >/= 18 to </= 80 years of age;
* Carotid stenosis (either symptomatic or asymptomatic);
* Planned carotid endarterectomy;
* Female patients must be non-pregnant and willing to use effective, redundant methods of contraception (i.e., for both self and male partner) throughout the study and for at least 30 days after discontinuation of study drug treatment;
* Male patients must agree to use a medically acceptable contraceptive (abstinence or use of a condom with spermicide) throughout the study and for at least 30 days after discontinuation of study drug treatment;
* All patients must be capable of understanding and complying with the protocol and must have signed the informed consent document.

Exclusion Criteria:

* Lack of acoustic window allowing TCD recordings;
* Unable or unwilling to consent;
* Metallic prosthetic cardiac valve;
* Recent (<4 weeks) ischemic stroke involving >1/3 of the MCA territory;
* Any history of hemorrhagic stroke;
* Thrombocytopenia;
* Coagulopathy;
* Trauma or surgery within preceding 30 days;
* History of bleeding disorder, gastrointestinal ulcers, or other medical problem associated with an increased risk of bleeding;
* Use of warfarin and any chronic antithrombotic therapy other than acetylsalicylic acid and/or dipyridamole; patients previously treated with warfarin are eligible if the drug has been discontinued and the INR prior to randomization has returned to <1.3;
* Use of clopidogrel, unless it has been discontinued at least 5 days prior to randomization;
* Fibrinolytic or GPIIb/IIIa inhibitor treatment within the preceding 24 hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of ARC1779 Injection on the number of microembolic signals detected by transcranial Doppler (TCD) in the immediate postoperative period | Immediate Post-Operative Period
To evaluate the safety of ARC1779 Injection with respect to bleeding risk in patients in the perioperative period. | Perioperative Period

SECONDARY OUTCOMES:
To determine the effect of ARC1779 on the incidence of new ischemic lesions detectable with diffusion-weighted magnetic resonance imaging (MRI) after carotid endarterectomy | Up to 7 Days
To determine the general safety and tolerability of ARC1779 Injection in this surgical population | Up to 7 Days
To assess laboratory parameters related to ARC1779 pharmacokinetics (PK) and pharmacodynamics (PD) | Up to 7 Days
To assess the relationships among ARC1779 PD, PK, and the frequency of cerebral microembolism | Up to 7 Days
To assess the relationships among ARC1779 PD, PK, and safety parameters. | Up to 7 Days

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Markus, MD, Principal Investigator — St George's, University of London
Locations (7):
- United States (2):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Eddy Scurlock Stroke Center - Methodist Hospital, Houston, Texas
- United Kingdom (5):
  - Addenbrooke's Hospital, Department of Vascular Surgery, Cambridge
  - University Hospitals Coventry and Warwickshire NHS TRUST, Coventry
  - Leeds General Infirmary, Leeds
  - St. George's, University of London, Cranmer Terrace, London
  - University Hospital of South Manchester, Wythenshawe Hospital, Southmoor Road, Manchester

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581
- [Derived] Markus HS, McCollum C, Imray C, Goulder MA, Gilbert J, King A. The von Willebrand inhibitor ARC1779 reduces cerebral embolization after carotid endarterectomy: a randomized trial. Stroke. 2011 Aug;42(8):2149-53. doi: 10.1161/STROKEAHA.111.616649. Epub 2011 Jun 23. PMID 21700934